CLINICAL TRIAL: NCT05366283
Title: Single Ascending Dose and Repeat Dose Study to Evaluate Pharmacokinetics, Pharmacodynamics, and Safety of Sargramostim Administered Subcutaneously, by Intravenous Infusion, or by Inhalation in Healthy Adult Subjects
Brief Title: Study to Evaluate Pharmacokinetics, Pharmacodynamics, and Safety of Sargramostim Administered Subcutaneously, Intravenously, or by Inhalation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Partner Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PTX-001-005
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-05

CONDITIONS: Drug Kinetics; Drug Effects on Physiology
MeSH Terms: interventions — sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Cohort 1 (Part 1) (Experimental): Single dose of 250 microgram (mcg) sargramostim IV over 2 hours
  Interventions: Biological: sargramostim
- Cohort 2 (Part 1) (Experimental): Single dose of 25 mcg sargramostim SC
  Interventions: Biological: sargramostim
- Cohort 3 (Part 1) (Experimental): Single dose of 125 mcg sargramostim SC
  Interventions: Biological: sargramostim
- Cohort 4 (Part 1) (Experimental): Single dose of 250 mcg sargramostim SC
  Interventions: Biological: sargramostim
- Cohort 5 (Part 1) (Experimental): Single dose of 500 mcg sargramostim SC
  Interventions: Biological: sargramostim
- Cohort 6 (Part 1) (Experimental): Single dose of 250 mcg sargramostim IH
  Interventions: Biological: sargramostim
- Cohort 7 (Part 2) (Experimental): Two doses of 500 mg sargramostim SC, weekly
  Interventions: Biological: sargramostim

INTERVENTIONS:
Biological: sargramostim — Sargramostim is a glycosylated, yeast-derived recombinant human granulocyte-macrophage colony-stimulating factor.
  Other Names: Leukine®; rhu-GM-CSF

SUMMARY:
This single center, single ascending dose (SAD) and repeat dose study in healthy adults comprises 2 parts. Part 1 will consist of 6 SAD cohorts, in which different dose levels of sargramostim will be given by intravenous (IV) infusion, subcutaneous (SC) injection, or inhalation (IH) administration. Part 2 will consist of 1 repeat dose cohort in which sargramostim will begiven by SC administration.

Blood samples for PK assessment will be collected before and over 24 hours after each study drug administration. Blood samples for PD assessment will be collected before and up to 14 days after drug administration in Part 1, as well as before the first and up to 14 days after the second drug administration in Part 2. Safety and tolerability will be assessed throughout the study. For Cohort 5 of Part 1 only, 3 subjects will provide a CSF sample for PK assessmen tonce after SC drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female participants
* Nonsmoker or ex-smoker
* Able to provide informed consent and comply with all study procedures
* Body Mass Index within 18.5-30.0 kilograms/meter squared, inclusive
* Females of childbearing potential willing to use highly-effective method of birth control.

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* History of allergic to sargramostim or its excipients, other human GM-CSFs, or other yeast-derived products.
* History of severe allergic reactions to other drugs.
* History of or any current medical condition or laboratory finding that may jeopardize completion of the study, present an increased risk to the subject, or compromise interpretation of the study. .
* Immunization with COVID-19 vaccine within 14 days of the study.
* Scheduled immunization with COVID-19 vaccine during the study
* Use of prescription drugs within 28 days of the study or requirement for maintenance drugs during the study.
* Participation in another investigational drug study within 28 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
maximum concentration | Blood samples collected up to 24 hours post dose
time to maximum | Blood samples collected up to 24 hours post dose
Area under the concentration-time curve (AUC) from time 0 to 24 hours | Blood samples collected up to 24 hours post dose
AUC from time 0 to infinity | Blood samples collected up to 24 hours post dose
AUC from time 0 to 24 hours/infinity | Blood samples collected up to 24 hours post dose
Elimination half-life | Blood samples collected up to 24 hours post dose
Clearance | Blood samples collected up to 24 hours post dose
Steady state volume of distribution (IV administration only) | Blood samples collected up to 24 hours post dose

SECONDARY OUTCOMES:
Number of subjects with adverse events in Part 1 | Up to Day 15 in Part 1
Number of subjects with adverse events in Part 2 | Up to Day 22 in Part 2
Ratio of T-regulatory cells to T-effector cells in the blood. | Up to Day 15 in Part 1, up to Day 22 in Part 2
CD14/CD16/human leukocyte antigen-DR isotype (HLA-DR) absolute cell count | Up to Day 15 in Part 1, up to Day 22 in Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Ila Joshi, PhD, Study Director — Partner Therapeutics, Inc.
Locations (1):
- AltaSciences, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No